CLINICAL TRIAL: NCT07032922
Title: Exploring How to Adapt an Evidence-Based Mindful Self-Compassion Program for Young Adults With Li-Fraumeni Syndrome
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002467; 002467-C
Record Dates: First submitted 2025-06-19; First posted 2025-06-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12-08

CONDITIONS: Li-Fraumeni Syndrome
Keywords: Li-Fraumeni Syndrome; Mindful Self-Compassion (MSC); Young Adults; LFS; MSC; Mental Health
MeSH Terms: conditions — Li-Fraumeni Syndrome; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stakeholders: Other key stakeholders (non-YAs, non-NIH researchers), such as LFS clinicians, advocacy group representatives, and researchers will be referred by colleagues. Our goal is to enroll a minimum of 3 and a maximum of 6 individuals who have different LFS expertise (e.g., genetics providers, psychosocial researchers, LFS community leaders) to capture diverse viewpoints important to adaptation of evidence-based interventions.
- YAs with LFS: Young Adults (18 up to 29 years old) who have been diagnosed with Li-Fraumeni Syndrome, half of whom have a cancer history and half of whom have no cancer history.

SUMMARY:
Background:

Li-Fraumeni syndrome (LFS) is a genetic disorder that increases the risk of cancer. People who have LFS are 24 times more likely to develop cancer than those who do not. Past research studies have shown that living with high cancer risk can cause distress in young adults with LFS. Mindful self-compassion (MSC) is a therapeutic resource that has helped people with and without cancer cope with distress and other mental health challenges. Researchers at the National Cancer Institute (NCI) want to know if an MSC program can be adapted for young adults with LFS.

Objective:

Demonstrate and get feedback on an MSC resource for young adults with LFS.

Eligibility:

Young adults aged 18 to 29 years with LFS who have not participated in an MSC program in the past 6 months and who do not participate in daily meditation for 30 minutes or more. Individuals must be willing to travel to the National Cancer Institute for a one-day demonstration.

Design:

Participants will answer a short online questionnaire to determine study eligibility, which may include questions about cancer history and mental health. Eligible participants will attend an in-person demonstration of the MSC resource. A small group of other people, such as health care providers, may also attend. Participants will be invited to give their feedback on the MSC resource and discuss how to make it relevant and helpful for young adults with LFS.

The demonstration will be held at the NCI campus in Rockville, Maryland. If the demonstration cannot be held in person, it will be conducted virtually. The total time to participate will be about 5.5 hours.

DETAILED DESCRIPTION:
Study Description:

Young adults (YAs) with Li-Fraumeni syndrome (LFS) often experience high levels of distress and complex and dynamic health burdens. Evidence-based interventions that might ameliorate these challenges, such as a mindful self-compassion (MSC) program, have not been tested for acceptability and appropriateness among YAs with LFS. The aim of this study is to determine how to adapt an evidence based MSC program to meet the needs and preferences of this population. Data from this study will inform the development of an adapted MSC intervention to address a significant gap in LFS supportive care for YAs.

Objectives:

The primary objective of this study is to convene YAs with LFS and other key stakeholders (e.g., LFS clinicians) at the National Cancer Institute (NCI) to demonstrate core components of an evidence-based MSC program and obtain feedback on how to adapt the program for YAs with LFS.

Endpoints:

This is a descriptive study; therefore, we are not generating a priori hypotheses or measuring outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, YAs must meet all of the following criteria:

* Self-reported diagnosis of LFS.
* Aged 18 to 29 years at the time of enrollment.
* Ability to speak, read, and/or write in English (to understand and provide informed consent and participate in the study activities).
* Currently live in the U.S.
* Willing to engage in a demonstration of a mental health resource for YAs with LFS and provide feedback on it.
* Able to travel to the NCI Shady Grove Campus.
* Access to a computer, high-speed internet, and a webcam, which may be necessary if the study team cannot conduct the study at the NCI due to unforeseen circumstances (e.g., government policy, weather).
* Have not participated in a mindfulness- or compassion-based program within the past 6 months.
* Do not have a consistent meditation practice >= 30 minutes per day.

Eligibility based on these inclusion criteria will be determined via an online screening questionnaire. To be eligible to participate in this study, non- YA stakeholders must meet all of the following criteria:

* At least age 18 at the time of enrollment.
* Ability to speak, read, and/or write in English (to understand and provide informed consent and participate in the study activities).
* Currently live in the U.S.
* Willing to observe a demonstration of a mental health resource for YAs with LFS and provide feedback on it.
* Able to travel to the NCI Shady Grove Campus.
* Access to a computer, high-speed internet, and a webcam, which may be necessary if the study team cannot conduct the study at the NCI due to unforeseen circumstances (e.g., government policy, weather).

EXCLUSION CRITERIA:

A YA who meets the following criteria will be excluded from participation in this study:

* A Patient Health Questionnaire (PHQ-9) score or a General Anxiety Disorder (GAD-7) score >= 15 at the time of screening. Scores >= 15 correspond to moderately severe or severe depression and severe anxiety, respectively. The PHQ-9 and GAD-7 are standardized, validated measures of depression and anxiety. The data obtained from participants who are determined to be ineligible will not be retained in the database or system. Instead, it will be destroyed to ensure the privacy and confidentiality of the participants.
* Individuals who do not meet eligibility criteria listed.

A non-YA stakeholder who meets any of the following criteria will be excluded from participation in this study:

-Individuals who do not meet eligibility criteria listed. No other exclusionary criteria apply.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will enroll up to 14 Young Adults with Li-Fraumeni Syndrome and up to 6 key stakeholders.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
To convene YAs with LFS and other key stakeholders to demonstrate core components of an evidence-based MSC program and obtain feedback on how to adapt the program for YAs with LFS | End of the study

CONTACTS AND LOCATIONS:
Overall Officials: Payal P Khincha, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- NCI Shady Grove Campus, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
For privacy issues data will only be shared as aggregate data after publication of results.